CLINICAL TRIAL: NCT02766933
Title: Cameroon Baptist Convention Health Board Chronic Hepatitis B Cohort Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Cameroon Baptist Convention Health (Other)
Responsible Party: Principal Investigator, Lewis R. Roberts, Principal Investigator, Mayo Clinic
Other Study IDs: 16-001716
Record Dates: First submitted 2016-04-20; First posted 2016-05-10 (Estimated); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis B; Hepatitis B, Chronic
Keywords: tenofovir; hepatocellular carcinoma; cirrhosis
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic; Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Serum and urine at enrollment and follow-up visits
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- hepatitis B cohort: CBCHB employees and/or spouses found to be hepatitis B surface antigen positive on screening

SUMMARY:
The natural history and response to therapy of chronic hepatitis B infection in West Africa are currently poorly understood. In this study, employees of the Cameroon Baptist Convention Health Board (CBCHB) and spouses who are found to be hepatitis B positive on screening will be offered enrollment. Disease monitoring and treatment will be provided following current WHO guidelines. Clinical data will be prospectively recorded for 5 years, and bio-specimens will be frozen for future analysis.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) is common in Cameroon, and hepatitis B-related hepatocellular carcinoma is a leading cause of cancer death throughout West and Central Africa. Little is known about the natural history of CHB in sub-Saharan Africa and the long term response to antiviral therapy. The study hypothesis is that these can be determined by prospective follow-up of a population-based cohort.

Aims, purpose, or objectives:

1. To determine the characteristics of a population of asymptomatic Cameroonian adults who work for the Cameroon Baptist Convention Health Board (CBCHB) who have chronic hepatitis B infection.
2. To determine the phase of infection into which these Hepatitis B carriers fall.
3. To determine the incidence and risk factors for cirrhosis, decompensated cirrhosis, and hepatocellular carcinoma in this cohort over time.
4. To offer treatment according to a standardized protocol, and to determine the outcome of treatment.
5. To archive serum samples from patients for potential future studies of specific markers associated with hepatitis B and liver disease outcomes.

Methods: Adult employees of the Cameroon Baptist Convention Health Board (CBCHB) and their spouses who are known to be positive for hepatitis B surface antigen (HBsAg+) will be offered the enrollment in a cohort study for CHB. Following enrollment, their stage of disease will be determined using clinical, laboratory and imaging studies. Patients will then be followed at regular intervals for 5 years. Antiviral therapy will be offered to patients who qualify according to current World Health Organization guidelines.

Significance: This protocol will prospectively determine the scope of CHB-related illness in an initially asymptomatic, population-based cohort and the outcomes of current WHO treatment guidelines in this African cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18yrs.
* CBCHB employee or spouse of an employee.
* Able to provide written informed consent.
* Willing to comply with follow-up visits.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CBCHB employees and their spouses who are found to be hepatitis B surface antigen positive during screening.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2016-05; Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each phase of chronic hepatitis B infection at enrollment | Enrollment
  distribution of subjects across the 4 phases of chronic hepatitis B at enrollment (immune tolerant, immune clearance, inactive carrier, and reactivation phases). This is determined by enrollment age, ALT, HBeAg status, clinical and imaging findings of cirrhosis, and (in some cases) serum hepatitis B DNA quantification
yearly incidence of compensated and decompensated cirrhosis in the study cohort | 5 years
  incidence of compensated and decompensated cirrhosis over time in the study cohort, as determined by interval history, physical exam, APRI (AST to platelet ratio index), and ultrasound findings
yearly incidence of hepatocellular carcinoma in the study cohort | 5 years
  incidence of hepatocellular carcinoma over time in the study cohort as determined by serum alpha fetoprotein, per-protocol imaging studies, and biopsy when appropriate
Percentage of treated subjects who achieve and maintain a complete response to antiviral treatment. | 5 years
  Percentage of subjects receiving antiviral treatment who achieve and maintain a complete response as determined by normalization of serum transaminases and (in some cases) loss of detectable serum hepatitis B DNA

CONTACTS AND LOCATIONS:
Overall Officials: Norah Nyah, M.D., Principal Investigator — Cameroon Baptist Convention Health Board
Locations (1):
- Mbingo Baptist Hospital, Bamenda, Northwest, Cameroon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials